CLINICAL TRIAL: NCT06259136
Title: Palliative Care Yields Cancer Wellbeing Support
Acronym: Pal-Cycles
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Collaborators: Lancaster University (Other); University Hospital, Bonn (Other); University of Navarra (Other); University in Zielona Góra (Other); University of Pecs (Other); European Association for Palliative Care (EAPC) (Unknown); Universidade Católica Portuguesa (Other); Hospice Villa Speranza (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Health Services Research
Other Study IDs: 101057243
Record Dates: First submitted 2024-02-06; First posted 2024-02-14 (Actual); Last update posted 2025-07-28 (Actual); Status verified 2025-03

CONDITIONS: Cancer
Keywords: Palliative care; Transitional care; End of life care
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Intervention Model Description: For this study a cross-sectional stepped wedge clustered clinical trial will be conducted.
  The design will start by an initial period in which all clusters e.g. different hospital sites, are part of the control group in which the patients receive care as usual. Subsequently, groups of clusters are exposed to the intervention at regular intervals (steps) until all clusters patients in all clusters have received care as defined in the intervention. The decision about which group of clusters will receive the intervention at which point in time is decided by randomization
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pal-Cycles Intervention (Experimental): The patients in the intervention arm will be exposed to the Pal-Cycles intervention.
  Interventions: Procedure: A transitional palliative care intervention
- Care as usual (No Intervention): The patients included in this intervention will be given care as usual.

INTERVENTIONS:
Procedure: A transitional palliative care intervention — The Pal-Cycles intervention starts just before the care transition from curative oncology care to palliative care with a goals of care conversation between a hospital care provider and the patient. The conversation will be recorded in a summary of treatment and care form which will be completed by a hospital based clinician based on the key elements of the conversation with the patient and the treatment and care plan. Afterwards a (digital) copy of the form is given to the patient and another copy is sent to the general practitioner in combination with the discharge letter.
  Other Names: Pal-Cycles intervention
  Arms: Pal-Cycles Intervention

SUMMARY:
The goal of this study is to evaluate the effectiveness of a programme for transitional palliative cancer care (Pal-Cycles) in seven countries (the Netherlands, Germany, United Kingdom, Hungary, Poland, Romania and Portugal) and its consequent effects on the number of readmissions into hospital.

The main hypothesis for the study is: that fewer people in the intervention arm of the study will require hospital re admission than those having usual care.

Participants will be asked to fill in questionnaires regarding their quality of care and quality of life.

DETAILED DESCRIPTION:
The study described in this protocol, a stepped wedge clinical trial, is part of a larger research project named: The Palliative Care Yields Cancer Wellbeing Support Programme (Pal-Cycles). The aim is to test and evaluate the implementation of the Pal-Cycles intervention, by implementing it in 14 care setting across seven European countries (the Netherlands, Germany, United Kingdom, Poland, Hungary, Romania and Portugal.) The primary focus of the evaluation will be on measuring the effect of the Pal Cycles intervention using the number of patients being readmitted into hospital after they had transferred to community care in comparison with patients receiving usual care. Additional relevant outcomes will also be gathered and analysed such as: the patient's quality of life, the experience from the family carer and the experience from the healthcare professional. Finally, an economic analysis will be embedded in the stepped wedge design.

The goals of the overarching research project are as follows:

1. To develop, implement and evaluate a transitional palliative cancer care intervention, with an intervention (the Pal-Cycles intervention) that aims for a smooth transition from the hospital to community-based care in the final months of life.
2. Adaptation of the transitional palliative cancer care intervention for patients with advanced cancer for its implementation in seven European countries within the project.
3. Training of oncologists in identifying patients with palliative care needs, establishing collaboratively comprehensive treatment and care plans, delivering patient-centred communication around discharge planning, advance care planning, and end-of-life care.
4. A clinical trial using a stepped wedge design will be implemented in fourteen care settingsacross seven European countries.
5. An implementation support intervention will guide the implementation of the clinical trial in all settings and will investigate barriers and opportunities for implementation and provide tailormade solutions where needed.
6. Dissemination of project results.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 years or above
* Patients diagnosed with advanced cancer
* Patients that are expected to develop or already may have palliative care needs
* Patients who are in transition from curative (hospital) to palliative care (community care)

Exclusion Criteria:

* People with cancer unable or unwilling to provide consent to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1050 (Estimated)
Dates: Start 2024-06-01 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2027-08 (Estimated)

PRIMARY OUTCOMES:
The difference in number of readmissions into hospital between the patients in the intervention arm and controle arm | 90 days after the end of the study or after death.
  The primary outcome of this research project will be the difference between the readmission rate from the control group and the intervention group. This was chosen based on the presumption that if the communication between healthcare professionals improves, the transition to home will be better and patients will be less likely to require hospital care. Another advantage is that it is a feasible and often well documented outcome measure which can be retrieved across multiple sites in multiple countries. A second advantage especially relevant for studies concerned with palliative care patients is that it can be measured early, as many patients die (of unrelated causes) during the study. By measuring early measurement compliance can be ensured.

SECONDARY OUTCOMES:
Demographic characteristics relative | 14 days after baseline.
  In order to gain some background on which relative is filling in the FAMCARE, the relative will also be asked some demographic questions concerning their age, gender and relationship to patient.
European Organization for Research and Treatment for Cancer Quality of Life Questionnaire C30 | Baseline, 30 days and 90 days after baseline.
  In addition to the number of admissions, another important indicator for the effectiveness of the Pal-Cycles interventions is the quality of life of life. To measure this multiple questionnaires will be used. One of them being the EORTC QLQ-C30. The questionnaire comprises of 30 questions assessing the patients ability to function from a physical, emotional, cognitive and functional point of view. For 28 of the questions the response can be given via a four point Likert scale giving the options: not at all, a little, quite a bit, very much. Where 1, not at all, indicates a higher score than 4, very much. The last two questions can be responded to via a visual analogue scale from 1 to7 (poor to excellent). Where 7, excellent, indicates a higher score than than 1, poor.
The Functional Assessment of Cancer Therapy - General (FACT-G) | Baseline, 30 days and 90 days after baseline.
  The other questionnaire that will be used to measure the patients quality of life is the FACT-G. The FACT-G was specifically developed to measure the cancer patient's health-related quality of life. This questionnaire for current and former cancer patients, is made up of 27 questions regarding quality of life by assessing wellbeing in four domains: physical, emotional, cognitive and functional. To all questions can be responded by filling in a 5 point likert scale; not at all, a little bit, somewhat, quite a bit and very much. Where 0, not at all, indicates a better score than 4, very much.
The Consultation and Rational Empathy measure (The CARE measure) | 14 days after baseline
  Another important outcome measure for this study is whether or not the Pal-Cycles intervention improves the quality of care. A key part of the Pal-Cycles intervention is the conversation between the clinician and the patient where the transition from curative oncological care to palliative care is discussed. To evaluate this conversation the CARE measure was included in the study. This questionnaire consists of ten Likert scale questions in which the emotional, ethical, cognitive and behavioural elements of the consultation.
  The patients can respond to the questionnaire by using a five point Likert scale consisting of the following options: 1 poor,2 fair, good,3 very good, 4 excellent. Where 4 excellent is indicating a better conversation than 3 very good.
Caregiver Network Analysis | 30 days after baseline
  The Caregiver Network Analysis was developed based on existing literature during a previous European project Insup-c for the purposes of a care network analysis. In the current project the objective is to improve the transition from curative care at the hospital to palliative care at home by ameliorating the communication between healthcare professionals. The questionnaire could assist in establishing if this is effective. The caregiver network analysis consists of twelve questions about which healthcare providers the patient has contact with as well as how the patient perceives their level of cooperation and quality of care. The answer options vary from dichotomous answer categories and open ended answers to 5- point Likert scales which have a range from 0 to 4. Where 4 , strongly agree, indicates a better score than 0 strongly disagree.
FAMCARE | 14 days after baseline
  Family carers play a large role in caring for patients with palliative care needs. There is an international trend to reduce hospital admission days and stimulate, community care, in order to decrease healthcare costs, but also to empower patients and their families. Therefore, measuring the family satisfaction with care has become integral to evaluating the quality of care. A scale that has proven to be a reliable measurement instrument is the FAMCARE. It was developed to measure satisfaction on performance of individual care takers performance of family members of patients with advanced cancer. This questionnaire consists of 20 questions to which can be responded to by a five point Likert scale. Where 1, very satisfied, indicates a better score than 5, very dissatisfied.
Place and date of death | 90 days after the end of the study or after death.
Presence of Advance decisions to refuse treatment (ADRTs) and Advance care plans (ACPs) as referred to in the hospital medical records. | 90 days after the end of the study or after death.
Referrals to palliative care services | 90 days after the end of the study or after death.
Economic analysis to assess the consequences of the intervention on health outcomes and resource utilization | 90 days after the end of the study or after death.
Demographic characteristics patients | Baseline.
  The demographic characteristics of the patient will be asked in a questionnaire. In addition to participating in the stepped wedge clinical trial described in this research protocol, they are also the co-lead on work package 5. This work package has as objective to analyse whether certain "sensitive" characteristics have influenced the quality of care of the patient during the oncology treatment. To limit patient burden the demographic characteristics in the questionnaire such as gender, age, civil status and members of the household will also be used as background information for the stepped wedge clinical trial.

CONTACTS AND LOCATIONS:
Overall Officials: Jeroen Hasselaar, Principal Investigator — Radboud University Medical Center (Radboudumc)
Locations (1):
- Radboudumc, Nijmegen, Gelderland, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
For WP3 the final dataset will be registered and deposited at the certified DANS-EASY archive. The data will be described with rich metadata in the English language.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: The data will be made available one year after the end of the study (2028) and will be available for 15 years.
Access Criteria: If applicants would like access to the datafiles they will need to ask permission from the access committee formed by Radboudumc and the principal investigator. This committee will weigh each request on its objectives. Requests will be sent to a mailbox of the Radboudumc, to guarantee accessibility with the then appointed employees.
URL: https://easy.dans.knaw.nl